CLINICAL TRIAL: NCT07049120
Title: Post-market Registry Study on the Safety and Efficacy of ZENFLEX Pro™ Peripheral Drug-eluting Stent System for Femoropopliteal Artery Lesions
Brief Title: Post-Market Study of ZENFLEX Pro Stent for Femoropopliteal Artery Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE-02
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZENFLEX Pro (Experimental): Subjects in this arm will receive treatment with the ZENFLEX Pro™ Peripheral Drug-eluting Stent System for femoropopliteal artery stenosis or occlusion. The procedure will be performed according to the device's instructions for use (IFU). Follow-up assessments will be conducted at 1, 6, and 12 months post-procedure to evaluate safety, efficacy, and performance outcomes.
  Interventions: Device: ZENFLEX Pro™ Peripheral Drug-eluting Stent System

INTERVENTIONS:
Device: ZENFLEX Pro™ Peripheral Drug-eluting Stent System — The ZENFLEX Pro™ Peripheral Drug-eluting Stent System will be implanted in patients with femoropopliteal artery lesions to evaluate safety and efficacy outcomes. The device is designed to provide mechanical support and deliver antiproliferative drug locally to reduce restenosis. The procedure will be performed via standard endovascular techniques.

SUMMARY:
This is a prospective, multi-center, single-arm post-market study evaluating the safety and effectiveness of the ZENFLEX Pro™ Drug-eluting Stent in treating femoropopliteal artery stenosis or occlusion. A total of 153 subjects will be followed at 1, 6, and 12 months. The primary endpoint is primary patency at 12 months.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm, post-market registry study designed to ensure continued evaluation of real-world safety, performance and efficacy of the ZENFLEX Pro™ Peripheral Drug-eluting Stent System in the treatment of femoropopliteal artery stenosis or occlusion. A total of 153 subjects will be enrolled in this study. Follow-up visits will be scheduled at 1-, 6-, and 12-months post-procedure. The primary endpoint is primary patency at 12 months. Secondary endpoints include technical success, procedural success, secondary patency rate, target lesion revascularization (TLR), clinically driven target lesion revascularization (CD-TLR), Rutherford classification, and ankle-brachial index (ABI). Safety endpoints include major adverse events, adverse events, all-cause mortality, major amputations, minor amputations, and stent fractures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion Criteria:

  1. Aged 18 to 80 years, regardless of gender.
  2. Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3, 4 or 5.
  3. Subject (or legal guardian, if applicable) is willing and able to provide consent before to the performance of any study-specific tests or procedures, has signed the consent form and agrees to attend all required follow-up visits.
* Angiographic Inclusion Criteria:

  1. Stenotic, restenotic or occlusive lesion(s) located in the native superficial femoral artery (SFA) and/or proximal popliteal artery (PPA) (i.e., within the P1 segment):

     1. Degree of stenosis ≥70% by visual angiographic assessment.
     2. Vessel diameter ≥4.0 mm and ≤6.5 mm.
     3. Total lesion length (or series of lesions) ≥ 10 mm and ≤ 140 mm (Note: Lesion segment(s) must be fully covered with one stent).
     4. Chronic total occlusion with a total lesion length of ≤120 mm.
  2. Patent popliteal and infrapopliteal arteries, with single-vessel runoff or better, defined as at least one of the three vessels remaining patent (i.e., <50% stenosis) down to the ankle or foot.

Exclusion Criteria:

* Clinical exclusion criteria:

  1. Pregnant or breastfeeding women, or women/men planning to conceive.
  2. Subjects who have had or are planned for major amputation (at or above the ankle level).
  3. Subjects known to be allergic or intolerant to materials used in the investigational device or treatment drugs, including nitinol, paclitaxel, aspirin, clopidogrel, heparin, rivaroxaban, contrast agents, etc.
  4. Subjects with serum creatinine ≥2.5 mg/dL or currently undergoing dialysis.
  5. Subjects with known, uncorrectable hemorrhagic disorders or severe coagulation dysfunction (prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≥2 times the upper limit of normal, or platelet count <80×10⁹/L).
  6. Previously stented target lesion/vessel.
  7. Target lesion/vessel previously treated with drug-coated balloon <12 months prior to enrollment.
  8. Subjects with a life expectancy of less than 1 year.
  9. Subjects who have received local or systemic thrombolysis treatment within 48 hours prior to enrollment.
  10. Subjects diagnosed with major clinical diseases or unstable conditions within the past 3 months, such as severe heart failure, unstable angina, myocardial infarction, transient ischemic attack or stroke, severe neurological or psychiatric history, severe infections, gastrointestinal bleeding, or active disseminated intravascular coagulation.
  11. Subjects currently participating in another clinical trial involving drugs or medical devices.
  12. Subjects whom the investigator considers unsuitable for participation in the clinical trial.
* Angiographic exclusion criteria:

  1. Presence of aneurysm in the target vessel.
  2. Heavily calcified lesions (Peripheral Arterial Calcium Scoring System [PACSS] grades 3-4).
  3. The target lesion requires the use of plaque excision, laser, or other debulking devices that may damage the vessel intima.
  4. The guidewire cannot pass through the target lesion, or percutaneous transluminal angioplasty (PTA) balloon cannot be used for pre-dilation.
  5. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reaching Primary Patency | 12 months post-procedure
  Primary patency is defined as a binary endpoint and will be determined to be a success when the duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) is ≤2.4 at the 12-month follow-up visit in the absence of clinically driven TLR or bypass of the target lesion.

SECONDARY OUTCOMES:
Number of participants with successful stent delivery and deployment resulting in ≤30% residual stenosis | During the procedure
  Technical success is defined as the delivery and deployment of the assigned study stent to the target lesion to achieve residual angiographic stenosis no greater than 30% assessed visually.
Number of participants with procedural success (technical success and no MAEs within 24 hours) | Within 24 hours post-procedure
  Procedural success is defined as technical success with no major adverse events (MAEs) noted within 24 hours of the index procedure.
Number of participants with primary patency | 6 months post-procedure
  Primary patency is defined as a binary endpoint and will be determined to be a success when the duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) is ≤2.4 at the 12-month follow-up visit in the absence of clinically driven TLR or bypass of the target lesion.
Number of participants with secondary patency | 6 and 12 months post-procedure
  Secondary patency at 6 months and 12 months. Secondary patency is defined as the absence of restenosis in the target lesion on DUS follow-up, with a diameter stenosis of ≤50% (PSVR ≤2.4), regardless of whether the target lesion has undergone reintervention.
Number of participants undergoing target lesion revascularization (TLR) | At 1, 6, and 12 months post-procedure
  TLR is defined as any repeat revascularization (endovascular or surgical) of the target lesion due to restenosis or occlusion, regardless of symptoms or diagnostic findings.
Clinically Driven Target Lesion Revascularization (CD-TLR) | At 1, 6, and 12 months post-procedure
  A target lesion revascularization will be considered clinically driven if it occurs within 5 mm proximal or distal to the original treatment segment with diameter stenosis ≥50% by quantitative angiography (QA) and the subject has recurrent symptoms (≥1 change in Rutherford Classification or associated with decreased ABI/TBI of ≥20% or ≥0.15 in the treated segment. TBI allowed in cases of incompressible vessels.)
Change in Rutherford Classification at 1, 6, and 12 months | 1, 6, and 12 months post-procedure
  Rutherford Peripheral Arterial Disease (PAD) Classification is a clinical grading system used to assess the severity of lower limb ischemia. The scale ranges from 0 to 6, where higher scores indicate more severe disease. Each category is defined by clinical symptoms and objective hemodynamic criteria as follows:
  0: Asymptomatic - Normal treadmill or stress test
  1. Mild claudication - Completes treadmill test; post-exercise ankle pressure (AP) <50 mmHg, and >25 mmHg drop from resting blood pressure
  2. Moderate claudication - Symptoms between categories 1 and 3
  3. Severe claudication - Cannot complete treadmill test; post-exercise AP <50 mmHg
  4. Ischemic rest pain - Resting AP <40 mmHg, with flat or low-amplitude ankle/metatarsal pulse volume recording (PVR); toe pressure (TP) <30 mmHg
  5. Minor tissue loss - Non-healing ulcer or localized gangrene with edema; resting AP <60 mmHg, ankle or metatarsal PVR flat or low amplitude; TP <40 mmHg
  6. Major tissue loss - Tissue loss extendi
Change in Ankle-Brachial Index (ABI) from baseline at 1, 6, and 12 months | 1, 6, and 12 months post-procedure
  The ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm as follows:
  Ankle: The systolic pressure will be measured in the target limb at the arteria dorsalis pedis and/or the arteria tibialis posterior. If both pressures are measured, the highest pressures will be used for the ABI calculation.
  Brachial: The systolic pressure will be measured in both arms, and the highest of both pressures will be used for the ABI calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Liu, Study Director — Zhejiang Zylox Medical Device Co., Ltd.
Locations (1):
- American Heart of Poland, Małopolskie Cardiovascular Center PAKS Chrzanów, Chrzanów, Chrzanów, Poland

IPD SHARING:
Plan to Share IPD: No